CLINICAL TRIAL: NCT06190353
Title: Development, Acceptability and Preliminary Efficacy of an Internet-Based Self-Help Program Using Acceptance and Commitment Therapy for Coping With Burnout Among Healthcare Workers: A Randomized Controlled Pilot Study
Brief Title: Development, Acceptability and Preliminary Efficacy of an Internet-Based Self-Help Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CanSagligi Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSV202301
Record Dates: First submitted 2023-12-07; First posted 2024-01-05 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Burnout, Professional
Keywords: Burnout; Acceptance and Commitment Therapy; Web-based Intervention; Healthcare Workers
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: a parallel two arms pilot randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The experimental group which will have an immediate access to web-based psychotherapy.
  Interventions: Behavioral: An internet-based self-help program with minimal telephone support utilizing Acceptance and Commitment Therapy for alleviating burnout among healthcare workers.
- Control (No Intervention): A wait-list control group which have one month delayed access to intervention program.

INTERVENTIONS:
Behavioral: An internet-based self-help program with minimal telephone support utilizing Acceptance and Commitment Therapy for alleviating burnout among healthcare workers. — An eight module self help program
  Arms: Intervention

SUMMARY:
This study aims to evaluate acceptability and initial effectiveness of an internet-based self-help program utilizing Acceptance and Commitment Therapy specifically for healthcare workers, intending to address burnout.

DETAILED DESCRIPTION:
This pilot study is a randomized controlled trial of two parallel groups. The study will comprise of an intervention and a wait-list control group. The intention of this study is to evaluate the acceptability and preliminary efficacy of an internet-based self-help program with minimal telephone support utilizing Acceptance and Commitment Therapy for alleviating burnout among healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Currently employed in the healthcare field as a doctor, nurse, technician, pharmacist or other healthcare profession for a minimum of six months.
* Proficiency in using computer and email.
* Experiencing symptoms of burnout related to the workplace.

Exclusion Criteria:

* Currently prescribed psychotropic medication.
* Currently undergoing psychotherapy.
* Presently experiencing thoughts of suicide or self-mutilation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Burnout Assessment Tool | At baseline and 4 weeks
  Burnout Assessment Tool is a validated measure which evaluates to what extend people experience burnout.
Valued Living Questionnaire (VLQ) | At baseline and 4 weeks
  VLQ is a validated measure and its aim is to evaluate valued living.

SECONDARY OUTCOMES:
Acceptance and Action Questionnaire-2 (AAQ-2) | At baseline and 4 weeks
  AAQ-2 is a measure aiming to evaluate experiential avoidance
System Usability Scale (SUS) | 4 weeks
  SUS aims to measure evaluations of participants about an internet based program.
Attendance rate | 4 weeks
  To evaluate feasibility, participants attendance rate to the program will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Nalbant, MD, Principal Investigator — CanSagligi Foundation Center for Contextual Behavioral Science
Locations (1):
- CanSagligi Foundation, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data would be available upon request